CLINICAL TRIAL: NCT07287306
Title: Effects of BLa80 and LRa05 on the Gut Microbiota Metabolite Profile of Healthy Individuals: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of BLa80 and LRa05 on the Gut Microbiota Metabolite Profile of Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20251120
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Each placebo stick contained 3 g of dextrin. Dosage: one stick per day.
  Interventions: Dietary Supplement: Placebo
- BLa80 (Experimental): Each probiotic stick contained dextrin and 2 × 10¹⁰ CFU BLa80. Dosage: one stick per day.
  Interventions: Dietary Supplement: BLa80
- LRa05 (Experimental): Each probiotic stick contained dextrin and 2 × 10¹⁰ CFU LRa05. Dosage: one stick per day.
  Interventions: Dietary Supplement: LRa05

INTERVENTIONS:
Dietary Supplement: Placebo — The experimental phase of this study will last 8 weeks and each subject will receive 3 follow-up visits (week 0, week 4, week 8).
  Arms: Placebo
Dietary Supplement: BLa80 — The experimental phase of this study will last 8 weeks and each subject will receive 3 follow-up visits (week 0, week 4, week 8).
  Arms: BLa80
Dietary Supplement: LRa05 — The experimental phase of this study will last 8 weeks and each subject will receive 3 follow-up visits (week 0, week 4, week 8).
  Arms: LRa05

SUMMARY:
Gut microbiota play a key role in polyphenol metabolism, participating in the breakdown of dietary components and producing various small molecule metabolites that affect human health. However, little is currently known about how gut microbes metabolize dietary compounds and produce bioactive metabolites. This study aims to use metabolomics to precisely identify food-derived metabolites in the blood to investigate whether probiotics (BLa80, LRa05) can enhance the breakdown of dietary components and improve their absorption and utilization in the human body.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 60 years;
2. Healthy individuals;
3. Participants must provide written informed consent.

Exclusion Criteria:

1. History of gastrointestinal surgery, other gastrointestinal diseases, metabolic disorders, immunodeficiency, hyperthyroidism, or cardiac or liver disease;
2. Use of immunosuppressants;
3. Pregnant or breastfeeding women;
4. Participants who have taken antibiotics or probiotics within the previous 3 months;
5. Planned surgery during the study period;
6. Patients with neurological disorders or psychiatric illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Serum metabolomic profiles measured by HPLC-MS/MS | Baseline (week 0), week 4, and week 8 post intervention
  Untargeted serum metabolomic profiling will be performed using high-performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) to assess changes in circulating metabolite concentrations over time.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospttal, Sun Yat-sen University, Guangzhou, Guangdong, China